CLINICAL TRIAL: NCT07290998
Title: A Safety Study of Intratumoral Diffusing Alpha Radiation Emitters for the Treatment of Locally Recurrent Prostate Cancer
Brief Title: Treatment of Locally Recurrent Prostate Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-PRST-05
Record Dates: First submitted 2025-12-01; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Recurrent Prostate Cancer; Locally Recurrent Prostate Cancer
Keywords: Alpha radiation; Prostate Cancer; Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT) — An intratumoral insertion of radioactive sources [Ra-224 containing stainless-steel 316LVM tubes- (Alpha DaRT seeds)]. The seeds release by recoil into the tumor short-lived alpha-emitting atoms

SUMMARY:
This is a multi-center clinical study enrolling up to 12 participants . The primary objective of the study is to evaluate the safety of Alpha DaRT for the treatment of locally recurrent prostate cancer . The secondary objectives of the study is to evaluate the efficacy of the Alpha DaRT sources in locally recurrent prostate cancer patients assessed by biochemical and clinical evaluation of disease progression as well as overall survival

DETAILED DESCRIPTION:
This study will be a prospective, interventional, open label, single arm, multiple center study to assess the safety efficacy of Alpha DaRT . Eligible patients with Locally Recurrent Prostate Cancer will be categorized into the study.

The "Diffusing Alpha-emitter Radiation Therapy (DaRT)", based on the interstitial intratumoral placement of an encapsulated Radium-224 source (3.7 days half-life), is described in this study. These sources release short-lived alpha-emitting atoms into the tumor microenvironment by recoil. DaRT seeds will be inserted into the tumor according to a pre-determined plan.The delivery of the DaRT Sources into the prostate tumor is done by using the Alpha DaRT Alpha Prostate Applicator.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically proven prostate adenocarcinoma
* Biochemical recurrence by the Phoenix definition (PSA nadir + 2 ng/mL) and confirmed by a pre-treatment biopsy.
* Patients eligible for focal salvage brachytherapy
* Clinical stage T1-T2 on relapse; unilateral extracapsular extension (T3a) on MRI permitted except posteriorly relative to the rectum
* Pre-salvage PSA level (rPSA) < 10 ng/ml
* Target lesion is technically amenable for Alpha DaRT sources implantation.
* Targetable lesion by either PSMA PET-CT according to PERCIST v1.0 OR by multiparametric MRI according RECIST v1.1 (Patients who were classified as stage II according to MRI)
* Lesion size ≤ 5 cm in the longest diameter
* ECOG Performance Status Scale 0 - 2
* Life expectancy is more than 6 months
* WBC ≥ 3500/µl, granulocyte ≥ 1500/µl
* Platelet count ≥60,000/µl
* Creatinine ≤1.9 mg/dL
* AST and ALT ≤ 2.5 X upper limit of normal (ULN)
* INR < 1.4 for patients not on Warfarin
* Age ≥ 40 years old
* Subjects are willing and able to sign an informed consent form
* Patients must agree to use adequate contraception (vasectomy or barrier method of birth control) for 3 months after DaRT insertion

Exclusion Criteria:

* Concomitant immunotherapy within the past 4 weeks.
* Patients with lymph node or metastatic disease
* Known hypersensitivity to any of the components of the treatment.
* Patients undergoing systemic immunosuppressive therapy excepting intermittent, brief use of systemic corticosteroids.
* Patients with prior surgery or low-dose-rate (LDR) brachytherapy as the primary treatment of their prostate cancer.
* [For Stage 1 of the study only] Patients with prior high-dose-rate (HDR) brachytherapy or stereotactic body radiation therapy (SBRT) as the primary treatment of their prostate cancer.
* Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months.
* Patients with uncontrolled intercurrent illnesses including, but not limited to an active infection requiring systemic therapy or a known psychiatric or substance abuse disorder(s) that would interfere with cooperation with the requirements of the trial or interfere with the study endpoints.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, low risk prostate cancer, or in situ cervical cancer.
* Patient requires treatment not specified in this protocol which may conflict with the endpoints of this study including evaluation of response or toxicity of DaRT.
* Patients do not agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry, for the duration of study participation, and for 3 months after DaRT insertion
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT.
* High probability of protocol non-compliance (in opinion of investigator).

Ages: 40 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Safety -Serious adverse events | From Day 0, Up to 3 years
  The primary safety endpoint is the overall incidence of device related serious adverse events (SAEs) over the duration of the trial

SECONDARY OUTCOMES:
To evaluate the efficacy of DaRT seeds according to blood tests | 12 month study, 2 years follow up ±1 month every 6 months.
  Biochemical relapse-free survival rate (where relapse is defined according to the Phoenix definition: increase in PSA ≥2 ng/mL above the nadir)
To evaluate the efficacy DaRT seeds according to Overall survival | once every 6 months for 2 years after final follow-up visit at 12 months
  Overall survival
To evaluate the efficacy of DaRT seeds according to Life Questionnaire- QLQ- PR25 | at day 0, 30 , 12 months and once every 6 months for 2 years
  Quality of life measure by the QLQ-PR25 questionnaire. The score is- 1-Not at all snd 4 is - Very much .
To evaluate the efficacy of DaRT seeds according to Life Questionnaire-IPSS | at day 0, 30 , 12 months and once every 6 months for 2 years
  Quality of life measure by the IPSS- International Prostate Symptom Score. The score is- 1 is not at all and 5 is almost always.
To evaluate the efficacy of DaRT seeds according to Life Questionnaire-SHIM | at day 0, 30 , 12 months and once every 6 months for 2 years
  Quality of life measure by the SHIM - Sexual Health Inventory for Men score, the score is - 1 - very low and 5 is- very high .

OTHER OUTCOMES:
To evaluate the efficacy of DaRT seeds according to clinical evaluation measured by Physical Examination and ECOG Performance status. | up to 3 years
  The secondary objective of the study is to evaluate the efficacy of the Alpha DaRT sources in locally recurrent prostate cancer patients assessed by clinical evaluation of the physician assessment and Performance status score cale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis, the score is from- 1- fully active and 5- Dead.
To evaluate the efficacy of DaRT seeds according to Disease progression measured by MRI / PSMA PET | Up to 3 years
  The secondary objective of the study is to evaluate the efficacy of the Alpha DaRT sources in locally recurrent prostate cancer patients assessed by Disease progression .

IPD SHARING:
Plan to Share IPD: No